CLINICAL TRIAL: NCT06807918
Title: Effects of Ketone Supplementation on Brain Energetics and Alcohol Consumption in Alcohol Use Disorder
Brief Title: Effects of Ketones on Brain Energetics and Alcohol Consumption in Alcohol Use Disorder
Acronym: KABA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 857493; 1R01AA031570-01A1 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-02-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder; Ketosis
Keywords: Alcohol Use Disorder; Ketosis; Ketone supplement; Magnetic Resonance Spectroscopy
MeSH Terms: conditions — Alcoholism; Ketosis | interventions — Magnetic Resonance Spectroscopy; Ethanol; Alcoholic Beverages

STUDY DESIGN:
Intervention Model Description: There are 6 study visits in this study, 2 MRI visits, 2 FDG PET/CT scan visits, and 2 alcohol bar lab visits. Participants will randomly receive the Kenetik or placebo beverage at the first MRI visit, FDG PET/CT visit, and alcohol bar lab visit, and then the other intervention at the other visit.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, and study staff assessing participant outcomes will all be blinded to the study intervention during the study. The placebo beverage will look and taste like Kenetik. The bottle labeling on the Kenetik and Placebo will look the same. A designated unblinded staff member will be assigned to manage the IP ordering, storage, accountability, and participant randomizations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone Supplement, Kenetik (Active Comparator): Kenetik: Ketone Drink supplement containing D-beta-hydroxybutyric acid and R-1,3 butanediol. D-beta-hydroxybutyric acid (C4H8O3) and 1,3 butanediol (C4H10O2). We will give 25 g of ketones 3 times. Once at an MRI visit, once at an FDG PET/CT scan visit, and once at an alcohol bar lab visit.
  Interventions: Other: magnetic resonance imaging scan; Other: fludeoxyglucose-18 positron emission tomography scan; Other: Alcohol bar lab
- Placebo Beverage (Placebo Comparator): Taste-matched placebo beverage is given 3 times. Once at an MRI visit, once at an FDG PET/CT scan visit, and once at an alcohol bar lab visit.
  Interventions: Other: magnetic resonance imaging scan; Other: fludeoxyglucose-18 positron emission tomography scan; Other: Alcohol bar lab
- Alcohol beverage (Experimental): The alcoholic beverage will be created by using a standard dose of 0.5g/kg 0.43 g/kg for men and women respectively (50% vodka), calculated to achieve a BrAC of about 0.050%. The alcoholic beverage will be given once at bar lab 1 and again at bar lab 2.
  Interventions: Dietary Supplement: Kenetik; Other: Placebo beverage

INTERVENTIONS:
Dietary Supplement: Kenetik — Drink a single dose of ketone supplement 25g, three times, randomly given at 1 of 2 MRI scan visits, 1 of 2 FDG PET/CT scan visits, and 1 of 2 alcohol bar lab visits.
  Other Names: D-Beta-hydroxybutyric acid and R-1,3 butanediol; Ketone supplement
  Arms: Alcohol beverage
Other: magnetic resonance imaging scan — Each subject will undergo 2 research MRI scan evaluations of the brain (up to 90 min.). The MRI is FDA-approved 7.0T Magentom Prisma scanner (Siemens Medical Solutions USA, Inc., Malvern, PA) with an approved radiofrequency head coil.
  Other Names: MRI scan
  Arms: Ketone Supplement, Kenetik; Placebo Beverage
Other: fludeoxyglucose-18 positron emission tomography scan — Each subject will undergo 2 FDG PET/CT scans. FDG is a positron emitting radiopharmaceutical. In addition to the radioactive FDG tracer, a low-dose CT of the chest is typically performed with the FDG PET/CT for the purpose of anatomical registration and attenuation correction of PET images. There are no separate diagnostic CT scans performed as part of this study.
  Other Names: FDG PET/CT scan
  Arms: Ketone Supplement, Kenetik; Placebo Beverage
Other: Alcohol bar lab — Each subject will undergo 2 alcohol bar labs. Subjects will drink about 2 ½ standard alcohol beverages, based on their weight to reach a breath alcohol level of 0.050%.
  Other Names: Alcoholic beverages
  Arms: Ketone Supplement, Kenetik; Placebo Beverage
Other: Placebo beverage — Drink a single dose of placebo beverage, that will look and taste the same as the ketone supplement. Subjects will recieve the beverage three times, randomly given at 1 of 2 MRI scan visits, 1 of 2 FDG PET/CT scan visits, and 1 of 2 alcohol bar lab visits, opisite of the Kenetik beverage.
  Arms: Alcohol beverage

SUMMARY:
This is a randomized, double-blind, crossover trial to evaluate the immediate effects of a nutritional ketone supplement, Kenotic compared to placebo on brain function and alcohol consumption in individuals with alcohol use disorder. Participants will complete 2 MRI scans, 2 FDG PET/CT scans, and 2 alcohol bar labs and will randomly receive Kenetik at one lab and the placebo at the next lab. During the bar labs participants will consume a dose of alcohol (based on weight), to bring their breath alcohol concentration to about 0.050%.

DETAILED DESCRIPTION:
The purpose of this research is to study how a nutritional ketone supplement, Kenetik may affect brain function and alcohol consumption in individuals with alcohol use disorder.

The study will use two types of imaging to see how the brain responds to Kenetik versus a placebo beverage. The study will use magnetic resonance imaging (MRI) and fludeoxyglucose-18 (FDG) positron emission tomography (PET) scans to study the brain. MRI scans use large magnets to create a magnetic field and radio waves to produce images of the brain. The FDG PET/CT scans use small amounts of a radioactive imaging drug, a special camera, and a computer to evaluate brain and tissue functions. FDG PET/CT scans are routinely done to evaluate brain and other organ diseases. The study will test brain functions at rest and while viewing pictures of alcohol. Participants will be asked to complete 2 MRI scans and 2 PET scans. Participants will randomly receive the Kenetik at 1 MRI scan and at 1 PET scan and will receive the placebo at the other MRI and PET scan visits.

The study will use two alcohol bar labs to study how Kenetik may affect alcohol consumption. Participants will randomly receive Kenetik on one of the visits, and the placebo beverage at the other visit. At each bar lab, Participants will be asked to drink alcohol beverages.

The study is double-blinded, which means that participants and the study staff running the study visits will not know at which visit participants will receive the Kenetik or placebo beverage.

Visit 1. Consent and Screening Visit (this will last ~4-5 hours)

Participants are asked not to eat or drink anything except water on the day of the screening session. A a meal will be proved during the visit. A breathalyzer test will be given to ensure that participants breath alcohol levels are 0.020 or lower and are sober and able to make a well-reasoned decision about whether or not to participate in the study.

The following will occur at the screening session, following signed consent:

* Demographic information, such as date of birth, age, biological sex, race, and ethnicity will be collected.
* Current information about address and contact information to into the University of Pennsylvania electronic medical record system.
* Provide a urine sample of about 30 mL (approximately 2 tablespoons) to be used for a drug screening test. Results from this testing are used for research purposes only. Participants will be informed of eligibility status after testing, but specific results will not be shared.
* Woman of childbearing potential, will be tested for pregnancy.
* Study personnel will measure vital signs (blood pressure and pulse), weight, and height. A doctor or nurse practitioner will do a brief physical exam.
* Staff will ask about any vision impairment or concerns about the ability to complete tasks or questionnaires on a computer.
* Staff will interview participants with a brief psychiatric structured interview called the 'MINI'. The interviews will ask about any current and past drug and alcohol use, depressed mood symptoms, as well as other psychiatric symptoms, including suicidal thinking.
* Participants will complete a brief mental ability test called the 'Shipley Institute of Living Scale'.
* Participants will complete a paper and pencil assessment or a short interview regarding alcohol and smoking history, behaviors, mood, and any drug or alcohol use. Additionally participants will be asked about any substance cravings or withdrawal symptoms.
* Participants will complete several psychological questionnaires related to substance use, cravings, risk behaviors, mental health, personality, depression and anxiety, and quality of sleep.
* Participants will complete questions about any medications, recreational drugs, or supplements they may be taking.
* Participants will complete a questionnaire about the presence of metal in their body to determine if it is safe to undergo an MRI.
* A small amount of blood (approximately 2.75 tablespoons) will be drawn for screening lab tests (a blood count and chemistry panel).
* Staff will perform an oral swab rapid HIV test. Staff will inform participants of the results and provide information about HIV. If the test is positive, study staff will draw a tablespoon of blood to conduct a confirmatory HIV blood test (i.e., to confirm the positive oral test). A clinician will discuss the results of this test. If the blood test is positive for HIV, staff will provide a referral for medical care and a copy of the test to provide to the doctor. Participants who tests positive for HIV will not be eligible to enroll in this study, because even without symptoms of HIV, the infection can make it impossible to read the MRI test results accurately.
* Participants will complete several computer-based tasks on a laptop that will be provided by the study team. These tasks will test the following brain cognition measures including visual memory, willingness to delay a reward offered, response time in reacting to specific information on the screen, verbal learning and memory, impulsiveness, and reaction time and accuracy when asked to match up a series of test pictures that are different shapes and colors. The computer tasks will take you about 50 minutes to complete.

After the screening visit, staff will call participants to confirm that the study is a good fit and schedule the rest of the study visits.

Visits 2 & 3. Alcohol Bar Lab visits (approximately 5 hrs.) The following will occur on the day of the two bar lab visits for participants. Participants will not to eat or drink anything except water after midnight the day before and on the day of the lab visit.

* A Breathalyzer test to measure breath alcohol concentration. Participants are required to have a 0.000% BrAC to continue with the visit. Staff will perform a finger stick to test glucose and BHB levels, using an instant-read point of care meter. Staff will provide the glucose level and what the reading means. Staff will take weight and vital signs.
* Staff will ask about recent use of drugs, alcohol, nicotine, and substance use and then ask for a urine sample. This will be used for a rapid urine drug test, and if the test is positive continued participation in the study will be reviewed by a study doctor. For woman of childbearing potential, a small amount of the urine will be used for a pregnancy test. The result of the pregnancy test must show not pregnant for to continue to participate in the study.
* Staff will provide a light meal and participants will complete some questionnaires.
* Staff will review the current list of medications and vitamins provided at the screening visit and ask if anything has changed
* Approximately 30 minutes after eating, participants will be asked to drink the Kenetik beverage or placebo beverage within 15 minutes. Neither participants nor our staff will know which beverage was received.
* Approximately 30 minutes after drinking the Kenetik or placebo beverage, participants will drink an alcoholic beverage based on weight, within 15 minutes. This drink will bring BrAC to approximately 0.050%. Staff will record the BrAC, and ask participants to complete the questionnaire as listed in the below table.
* Staff will ask about any side effects that may occur throughout the lab procedures.
* Alcohol bar lab (~2 hours) Approximately 1 hour after the first dose of alcohol, staff will provide chips that equal $24 and that can be used to purchase more alcoholic beverages (8 mini drinks in total). Participants can decide to keep the money or use it to buy more drinks. Participants are required to stay in the lab room for ~2.5 hours in total. They can watch videos and read magazines during these hours.
* After the meal, staff will check BrAC, BHB, and Glucose a final time. Ask about any side effects and staff will schedule the second lab visit. The second visit will occur at least 2 days after this visit and will follow the same procedures. Participants may leave once their BrAC is below 0.010.
* Table of Lab Visits Approximate study times Procedure 1:00 PM Arrive at CSA 1:00-1:30 PM BrAC1, weight, vital signs, urine sample, finger stick for BHB, and Glucose, review of medications currently taking, and review of alcohol and drug use since last visit 1:30-2:00 PM light meal, and questionnaires1 2:00-2:15 PM Drink Kenetik or placebo beverage 2:15-2:30 PM BRAC2, and questionnaires2 2:30-2:45 PM Alcohol administration 2:45 PM BrAC 3 3:00 PM BrAC 4 3:15 PM BrAC 5, and Finger stick for BHB, and Glucose Ask about 3:30 PM BrAC 6, 3 questionnaires, Bar lab: first tray of 4 alcoholic mini-drinks.

4:30 PM BrAC 7, 3 questionnaires, Bar lab: second tray of 4 alcoholic mini-drinks.

5:00 PM BrAC 8 5:30 PM BrAC 9, and Study Intervention questionnaire 5:50 PM Meal, finger stick for BHB, and Glucose 6:00 PM BrAC 10, meet with study clinician and leaves by Lyft when BRAC is <0.010% and Glucose returns to normal levels of > 70 mg/dl.

*Time in the above table may vary due to delays in start time of the lab visit.

Follow-up Visit (approximately 5 minutes): A follow-up phone call will occur the day after each lab visit and the following will occur:

• Staff will ask about any side effects that may have been experienced.

Visit 4 & 5. MRI Scan visits (approximately 2 hours)

On the day before the scan visits, participants will not drink any alcoholic beverages after 10 PM. Staff will provide participants with a snack after the scanning visit is complete.

On the day of the study visits the following will be done:

* Meet a study team member at the Perelman Center for Advanced Medicine and complete the following tests:
* A Breathalyzer test to measure breath alcohol concentration. A 0.000% BrAC is required to continue with the visit. Study personnel will measure vital signs (blood pressure and pulse), weight, and height. Participants will provide a urine sample for urine drug testing and urine pregnancy for woman of childbearing potential. A positive drug test result will be reviewed by the PI for continued participation in the study.
* Staff will ask about any changes in any of the medications or vitamins that was reported since the last visit. Staff will be asked about recent use of alcohol, drugs, and nicotine since the last visit.
* Participants will drink the Kenetik beverage or placebo beverage within 15 minutes. Neither participants nor our staff will know which beverage was received.
* Participants will receive a brain 7-Tesla MRI scan (~1.5 hours). An MRI is a type of scan that uses radio waves to take detailed pictures of the body. Participants lie on an MRI table where the technologist will place a receiver on the part of the body to be studied (brain). A blanket will be provided for comfort and earplugs since the MRI makes noises while it is scanning. Participants will still be able to hear some sound to ensure communication with the technologist and follow any direction given throughout the MRI scan. The technologist will slowly slide participants into the MRI magnet where radio waves will be transmitted.

  * Participants will fill out an MRI safety form.
  * Participants will remove any metal they may be wearing.
  * Staff will provide earplugs for the noise from the MRI scanner, and positioning on the imaging table with head in the scanner, held comfortably in a special head holder.
  * Staff will provide instructions not to move the head and to lie as still as possible during the scan (~ 90 minutes). There will be several scans, during which staff will obtain a structural image of the brain, and measure levels of ketones (energy in the brain), neurotransmitter GABA and glutamate, and NAD (a cofactor involved in energy metabolism).
* After the MRI visit is complete staff will provide a light snack and participants may leave. Staff will call the next day to inquire about any side effects of the MRI day scan.

Visit 6 & 7. PET Scanner Visits (this will last 3 hrs.)

Participants will be asked to not eat or drink anything except water ~8 hours before the PET scanning visits.

On the day of the study visits the following will be done:

Meet a study team member at the Hospital of the University of Pennsylvania and complete the following tests:

* A Breathalyzer test to measure breath alcohol concentration. Participants are required to have a 0.000% BrAC to continue with the visit. Staff will perform a finger stick to test blood glucose and BHB levels, using an instant-read point of care meter. Staff will let participants know their glucose level and what the reading means. Staff will take weight and vital signs.
* Staff will ask about recent use of drugs, alcohol, nicotine, and substance use and then ask participants to give a urine sample. This will be used for a rapid urine drug test, and if the test is positive continued participation in the study will be reviewed by a study doctor. If a woman of childbearing potential, a small amount of the urine will be used for a pregnancy test. The result of the pregnancy test must show not pregnant to continue to participate in the study.
* Trained staff will place two IVs into a vein in arms or hands to draw blood and give the FGD tracer. Staff will measure vital signs (blood pressure and pulse), weight, and height. Blood will be drawn from the IV at 5-time points for study measures and sent to the lab for research results. Staff will measure glucose and BHB levels using an instant-read point-of-care meter. Staff will provide the results of the glucose level.
* A list of current medications and vitamins will be reviewed. Participants will be asked about any changes in medications, dosage, or frequency of use of any medications or vitamins
* Participants will drink the Kenetik beverage or placebo beverage within 15 minutes. Neither participants nor our staff will know which beverage was received.
* Imaging of FDG is done with specialized cameras that can pick up the tiny radiation signals given off by the radiotracer and determine where the signals come from. In this way, we can form a picture of where the radiotracer goes after it is injected. The type of scan staff will perform is called a PET/CT scan, which uses a large doughnut-shaped detection device to provide a map of where radiotracers go in the body. Because this study is experimental, participants will not receive the results or feedback from study participation.

Participants will be asked to remove any metal objects before entering the scanner. The FDG tracer will be injected using the IV after positioned on the scanner, lying face up on the scanner table for about 1 hour, while the PET/CT machine collects imaging information over the body. Blood samples will be drawn before the injection and at 5 other time points during the scan. Approximately 45 mL (about 9 teaspoons) of blood will be collected during the scan. The blood will be used to measure radioactive counts and/or test how the tracer is being metabolized by the body.

Since this is experimental, the information the FDG PET/CT scans will not affect any medical care being received. The medical record will only include information that says a research PET/CT scan was performed, the experimental results of the scan will not be included . If there are unexpected findings on the CT portion of the scan that may affect medical care, staff will communicate these findings and what they mean. Images from the FDG PET/CT scans will be stored on our clinical imaging archive system of the University of Pennsylvania Health System, but will not be used for any clinical care.

• After completing the PET/CT scan participants will complete 2 questionnaires and perform a finger stick to test glucose level. Staff will provide the results and what they mean and then provide a snack. If glucose level is below 70 mg/dL, then staff with perform another finger stick to test glucose level 15 minutes after the snack was eaten.

Follow-up On the first business day following the study visits, study staff or a study doctor will call to ask about any changes to health and to ensure that not side effects from the Ketentik or the FDG PET/CT scan occurred.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-65 years old
2. Able to provide written informed consent
3. Meets current DSM-5 criteria for mild to moderate (established using MINI)
4. Average weekly alcohol consumption of at least 15 standard drinks over the past month before consent (self-report)
5. Not seeking treatment for AUD (self-report)

Exclusion Criteria:

1. Unwilling or unable to refrain from use of alcohol, within 24 hours of Alcohol Bar Lab, MRI and PET procedures (self-report, breathalyzer).
2. Use of psychoactive medications or medications that may affect study results (self-report, medical history).
3. Current DSM-5 diagnosis of a major psychiatric disorder (other than alcohol, Marijuana, and nicotine use disorders) that required hospitalization or daily medication in the past year.
4. Current significant alcohol withdrawal symptoms in the past 12 months that required medical treatment (self-report, medical history).
5. A current, clinically significant physical disease or abnormality on the basis of medical history, physical examination, or routine laboratory evaluation that could interfere with study participation or make it hazardous for the subject to do so (e.g., bleeding disorder, pancreatitis, epilepsy, liver disease, kidney disease, or diabetes as determined by history and clinical exam); ALAT or ASAT concentration greater than 3 times the upper limit of normal (ULN), or bilirubin above the ULN. (Note-abnormal laboratory tests during screening may be repeated once).
6. Current, major gastrointestinal (GI) diseases, such as: GERD, Crohn's disease, Irritable bowel syndrome, Ulcerative colitis, Celiac disease Diverticulitis, or other clinically significant physical disease that may interfere with the intake of the Ketone Supplement based on medical history, and evaluation of the Study Physician.
7. Clinically significant laboratory findings that could affect brain function (e.g., HIV+).
8. Head trauma with loss of consciousness for more than 30 minutes (self-report, medical history).
9. Pregnant or breast-feeding
10. Weight greater than 250lbs (Need to cap amount of alcohol give based on weight to individuals).
11. BMI greater than 35.
12. Self-reported claustrophobia.
13. Contraindications to MRI (e.g., metal in the body that cannot be removed and is not MRI compatible).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To examine the effects of a single dose of KS compared to placebo on brain glucose energetics | 90 minutes
  The primary outcome measure to be analyzed is a comparison of a single dose of KS versus placebo in AUD subjects in the amount of FDG uptake (CMRg metabolic rate of glucose) (mmol/L) levels in the brain.
To examine the effects of a single dose of KS compared to placebo on brain ketone energetics | 90 minutes
  The primary outcome measure to be analyzed is a comparison of a single dose of KS versus placebo in AUD subjects in the amount of FDG uptake BHB (beta-hydroxybutyrate) (mmol/L) levels in the brain.

SECONDARY OUTCOMES:
To determine the effects of KS compared to placebo on alcohol pharmacokinetics and subjective responses following an alcohol priming dose. | 3 hours
  The outcome measure to be analyzed is a comparison of breath ethanol levels (grams/210liters of breath) in response to a priming dose of alcohol following administration of KS vs. placebo.
To determine the effects of KS compared to placebo on alcohol consumption. | 2 hours
  The outcome measure to be analyzed is a comparison of the number of alcohol drinks consumed during the bar lab, following the administration of KS vs. placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Corinde Wiers, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Studies of Addiction, Philadelphia, Pennsylvania, United States